CLINICAL TRIAL: NCT00002565
Title: RANDOMIZED COMPARISON OF ALTERNATING TRIPLE THERAPY ("ATT") VERUS CHOP IN PATIENTS WITH INTERMEDIATE GRADE LYMPHOMAS AND IMMUNOBLASTIC LYMPHOMAS WITH INTERNATIONAL INDEX 2-5
Brief Title: Combination Chemotherapy in Treating Patients With Intermediate-Grade or Immunoblastic Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000063574; MDA-DM-94017; NCI-T94-0040D; DM94-017 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2004-06-30 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: stage I grade 3 follicular lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage II grade 3 follicular lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Bleomycin; VAP-cyclo protocol; Cisplatin; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Idarubicin; Ifosfamide; Mesna; Methylprednisolone; Mitoxantrone; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Sequential 4-, 5-, and 3-Drug Combination Chemotherapy. IdSHAP: IDA/CDDP/ARA-C/MePRDL; followed by BIdCOS: BLEO/IDA/CTX/VCR/MePRDL; followed by MINE: Mesna/IFF/DHAD/VP-16.
  Alternating triple therapy (ATT) of IdSHAP (idarubicin, cisplatin, cytarabine, methylprednisolone), BIdCOS (idarubicin, vincristine, bleomycin, cyclophosphamide, methylprednisolone), and MINE (mesna, ifosfamide, mitoxantrone, etoposide).
  Interventions: Biological: bleomycin sulfate; Drug: cisplatin; Drug: cyclophosphamide; Drug: cytarabine; Drug: etoposide; Drug: idarubicin; Drug: ifosfamide; Drug: mesna; Drug: methylprednisolone; Drug: mitoxantrone hydrochloride; Drug: vincristine sulfate
- Arm II (Experimental): 4-Drug Combination Chemotherapy. CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone): CTX/DOX/VCR/PRED.
  Interventions: Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: bleomycin sulfate
  Arms: Arm I
Drug: CHOP regimen
  Arms: Arm II
Drug: cisplatin
  Arms: Arm I
Drug: cyclophosphamide
Drug: cytarabine
  Arms: Arm I
Drug: doxorubicin hydrochloride
  Arms: Arm II
Drug: etoposide
  Arms: Arm I
Drug: idarubicin
  Arms: Arm I
Drug: ifosfamide
  Arms: Arm I
Drug: mesna
  Arms: Arm I
Drug: methylprednisolone
  Arms: Arm I
Drug: mitoxantrone hydrochloride
  Arms: Arm I
Drug: prednisone
  Arms: Arm II
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective for intermediate-grade or immunoblastic non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have intermediate-grade or immunoblastic non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare, in a randomized setting, the time to treatment failure and the survival of patients with poor-prognosis intermediate-grade or immunoblastic lymphoma treated with the standard regimen of CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone) versus the new alternating triple therapy (ATT) of IdSHAP (idarubicin, cisplatin, cytarabine, methylprednisolone), BIdCOS (idarubicin, vincristine, bleomycin, cyclophosphamide, methylprednisolone), and MINE (mesna, ifosfamide, mitoxantrone, etoposide).

II. Compare the complete response rate achieved with ATT versus standard CHOP.

III. Assess the feasibility of delivering full standard doses of chemotherapy to patients over 60 years of age who receive granulocyte colony stimulating factor support.

IV. Compare the predictive capability of the M.D. Anderson Tumor Score System versus the International Index System.

OUTLINE: Randomized study. The following acronyms are used: ARA-C Cytarabine, NSC-63878 BLEO Bleomycin, NSC-125066 CDDP Cisplatin, NSC-119875 CTX Cyclophosphamide, NSC-26271 DHAD Mitoxantrone, NSC-301739 DOX Doxorubicin, NSC-123127 G-CSF Granulocyte Colony-Stimulating Factor (source unspecified) IDA Idarubicin, NSC-256439 IFF Ifosfamide, NSC-109724 MePRDL Methylprednisolone succinate Mesna Mercaptoethane sulfonate, NSC-113891 PRED Prednisone, NSC-10023 VCR Vincristine, NSC-67574 VP-16 Etoposide, NSC-141540

Arm I: Sequential 4-, 5-, and 3-Drug Combination Chemotherapy. IdSHAP: IDA/CDDP/ARA-C/MePRDL; followed by BIdCOS: BLEO/IDA/CTX/VCR/MePRDL; followed by MINE: Mesna/IFF/DHAD/VP-16.

Arm II: 4-Drug Combination Chemotherapy. CHOP: CTX/DOX/VCR/PRED.

PROJECTED ACCRUAL: 218 evaluable patients will be accrued over approximately 31 months to this multicenter study. If either arm is significantly inferior at interim analyses after 31 and 60 treatment failures, consideration will be given to early closure.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated non-Hodgkin's lymphoma (NHL) of one of the following histologies: Diffuse large cell Follicular large non-cleaved cell Diffuse mixed cell Immunoblastic At least 2 of the following poor-prognosis factors required: Age over 60 Performance status greater than 1 Any elevation of LDH More than 1 extranodal site Ann Arbor stage III or IV T- and B-cell NHL eligible if meeting all above criteria No primary CNS lymphoma Brain involvement eligible if not primary

PATIENT CHARACTERISTICS: Age: Over 15 Performance status: Any status Hematopoietic: (unless secondary to tumor) Absolute granulocyte count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL Elevation secondary to tumor discussed with study chairman Renal: (unless secondary to tumor) Creatinine no greater than 1.5 mg/dL Cardiovascular: Left ventricular ejection fraction greater than 55% by echocardiography Pulmonary: No chronic obstructive or restrictive lung disease Pulmonary consultation required in cases of doubt Other: No HIV infection No prior malignancy with less than a 90% 5-year survival probability No patients unable or unlikely to adhere to treatment because of geographic, economic, emotional, or social factors No unwillingness to accept blood product transfusions or other supportive measures (e.g., antibiotics)

PRIOR CONCURRENT THERAPY: No prior therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1994-05-25 (Actual); Primary Completion 2007-02-05 (Actual); Study Completion 2007-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States
- Faculdade de Medicina do ABC, São Paulo, Brazil
- Clinica Alemana, Santiago, Chile